# Statistical Analysis Plan (SAP)

Study No. LMS-003

A Phase 3, Double-Blind, Placebo-Controlled, Randomized, Parallel-Group Study to Evaluate the Efficacy and Safety of Amifampridine Phosphate (3,4-Diaminopyridine Phosphate) in Patients with Lambert-Eaton Myasthenic Syndrome (LEMS)

Version 1.0

July 12, 2017

Prepared for Catalyst Pharmaceuticals, Inc. 355 Alhambra Circle, Suite 1250 Coral Gables, FL 33134

Prepared by
STATKING Clinical Services
759 Wessel Drive
Fairfield, OH 45014
513-858-2989
www.statkingclinical.com



**STATKING Clinical Services** 

# **Approval Page**

I agree to the format and content of this document.

Approved by:

Steven Miller, PhD **Date** 

**Chief Operating Officer and Chief Scientific Officer** 

Catalyst Pharmaceuticals, Inc. 355 Alhambra Circle, Suite 1250 Coral Gables, FL 33134

smiller@catalystpharma.com

**Authored by:** 

Date

Dennis Clason, PhD **Statistician** 

STATKING Clinical Services 759 Wessel Drive Fairfield, OH 45014 513-858-2989 ext. 313

dclason@statkingclinical.com

Approved by (internal review):

**Date** 

Lori Christman, PhD Statistician

**STATKING Clinical Services** 759 Wessel Drive Fairfield, OH 45014 513-858-2989 ext. 317 lori@statkingclinical.com

Approved by:

Clare Geiger, RN **Date** 

**Project Manager STATKING Clinical Services** 759 Wessel Drive Fairfield, OH 45014 513-858-2989 ext. 304

clare@statkingclinical.com

# **Revision History**

# **Table of Contents**

| 1.0 SYNOPSIS OF STUDY DESIGN PROCEDURES | 6 |
|------------------------------------------------------|----|
| 1.1 Design and Treatment | 6 |
| 1.2 Study Procedures | 6 |
| 1.3 Sample Size | 7 |
| 2.0 DATA ANALYSIS CONSIDERATIONS | 7 |
| 2.1 Types of Analyses | 7 |
| 2.2 Analysis Populations | 8 |
| 2.3 Missing Data Conventions | 8 |
| 2.4 Interim Analyses | 9 |
| 2.5 Study Center Considerations in the Data Analysis | 9 |
| 2.6 Documentation and Other Considerations | 9 |
| 3.0 ANALYSIS OF BASELINE SUBJECT CHARACTERISTICS | 9 |
| 4.0 ANALYSIS OF EFFICACY | 9 |
| 4.1 Description of Efficacy Variables | 9 |
| 4.2 Analysis of Efficacy Variables | 10 |
| 5.0 ANALYSIS OF SAFETY | 12 |
| 6.0 OTHER RELEVANT DATA ANALYSES/SUMMARIES | 13 |
| 6.1 Subject Completion | 13 |
| 6.2 Study Drug Administration and Compliance | 14 |
| 6.3 Patient Data Profiles | 14 |
| 7.0 LIST OF ANALYSIS TABLES, FIGURES AND LISTINGS | 15 |
| 8.0 REFERENCES | 18 |

| Statistical Analysis Plan | LMS-003 |
|---------------------------------------------------------|---------|
| APPENDIX A – TABLES, FIGURES AND LISTING SPECIFICATIONS | 19 |
| APPENDIX B – TABLE SHELLS | 21 |

# 1.0 Synopsis of Study Design Procedures

This study is a prospective, randomized, placebo-controlled, multicenter study to evaluate the efficacy and safety of amifampridine phosphate in subjects diagnosed with Lambert Eaton Myasthenic Syndrome (LEMS). The endpoint assessments of this Phase 3 study are as follows:

- Primary:
  - To assess the clinical efficacy of amifampridine phosphate compared with placebo in adults with LEMS, based on change of the co-primary endpoints Quantitative Myasthenia Gravis (QMG) Score and Subject Global Impression (SGI).
- Secondary:
  - Clinical Global Impression of Improvement (CGI-I)
- Exploratory:
  - Greater than 20% increase in the average time of 3 repetitions for Timed Up and Go test (3TUG)
  - Subject rating on change of most bothersome symptom for them.

# 1.1 Design and Treatment

Subjects will be randomized on Day 0 to either treatment group in a 1:1 ratio. Investigational product (IP) will be administered under double-blind conditions such that neither the Investigator nor subject knows if they are taking placebo or amifampridine phosphate.

Amifampridine phosphate (at the subject's optimal dose established prior to enrollment into this trial) or placebo will be dispensed by the site pharmacist, according to the randomization schedule, to begin with the next dose after all Day 0 assessments are completed and continued for 4 days. Although subjects at the high (dose  $\geq$  60 mg/day) and low (dose < 60 mg/day) are randomized separately, the study is not powered to detect differences across dose levels and no inferential analyses are planned to compare dose levels (See Section 1.3). The amifampridine phosphate dose is 30 mg to 80 mg total daily dose (expressed as freebase form), given in 3 to 4 divided doses, with no single dose >20 mg.

#### 1.2 Study Procedures

The planned duration of participation for each subject is 5 days (Day 0 through Day 4), excluding the screening period, which can last up to 7 days. Those subjects satisfying all inclusion and exclusion criteria will be randomized to a Treatment Group on the last day of the screening period (Day 0). The treatment period will take place on the remainder of Day 0 and Days 1 through 4. The following assessments will be performed at the beginning and end of the 4-day treatment period:

- Vital signs
- Urine sample for amifampridine level (collected at days 3, and 4)
- Clinical Global Impression of Improvement (CGI-I)
- Subject Global Impression (SGI)
- Quantitative Myasthenia Gravis (QMG)
- Triple Timed Up and Go (3TUG)
- Patient most bothersome symptom question
- Record concomitant medications
- Monitor for adverse events (throughout the 5-day treatment period)

# 1.3 Sample Size

The study is powered with respect to the co-primary efficacy endpoints of the study. For change from baseline (CFB) in QMG Scores, a between-treatment difference of -3.5 and a standard deviation of at most 3, a sample size of at least 24 subjects will provide power of at least 80% for a 0.05 level two-sided test. Similarly, for CFB in SGI Scores, a between-treatment difference of -2.1 and a standard deviation of at most 2, a sample size of at least 26 subjects will provide power of 80% for a 0.05 level two-sided test. Thus a total sample size of 26 subjects, equally randomized to two treatment sequences, will provide power of at least 80% for each of the two co-primary endpoints.

The randomization is stratified by high and low dose of the investigational product. Due to the fact that each dose strata has an insufficient number of observations to be adequately powered to do meaningful hypothesis testing, no statistical comparisons by treatment will be done for individual dose-strata subgroups.

# 2.0 Data Analysis Considerations

# 2.1 Types of Analyses

Analyses will consist of summarizing efficacy and safety data. Unless otherwise stated, two-sided P values <0.05 will be considered as statistically significant.

The following standards will be applied for the analyses unless otherwise specified. Simple summary statistics (descriptive statistics) for continuous data are: n (number of non-missing observations), mean, median, standard deviation, minimum, and maximum. The frequency count and percentage will be used to summarize categorical data. Summary statistics will be presented by treatment. All data collected will be presented in the by-subject data listings, sorted by subject and by time point, where appropriate.

Additionally, the randomization is stratified by high and low dose of the investigational product. Therefore, descriptive statistics, grouped by both

treatment and dose level strata, will be presented using the same descriptive analyses described above for continuous and categorical data, as applicable.

# 2.2 Analysis Populations

The following analysis populations will be defined:

**Safety:** This population consists of all randomized subjects who receive at least 1 dose of IP (amifampridine or placebo).

**Full Analysis Set (FAS), Intent to Treat Population:** This population consists of all randomized subjects who receive at least 1 dose of IP (amifampridine or placebo) and have at least one post-treatment efficacy assessment.

**Per Protocol (PP):** This population is a subset of the FAS population, excluding subjects with major protocol deviations. The PP population will include all subjects who:

- Have no major protocol deviations or inclusion/exclusion criteria deviations that might potentially affect efficacy, and
- Subjects who took at least 80% of the required treatment doses and remained enrolled for at least 4 days.

Evaluations obtained at the time of discontinuation will be included in the FAS and PP analyses, as applicable. Subjects who discontinue with no post-randomization data (no Day 0 and no Day 4 data) will be excluded from all efficacy analyses but will be included in the safety analyses.

Exclusion from the FAS and PP Populations will be finalized prior to database lock and subsequent unblinding.

# 2.2.1 Subgroup Definitions

Descriptive statistics for each efficacy variable will be provided by low dose (less than 60 mg/day) and high dose (60 mg/day, and higher) subgroups for subjects receiving amifampridine or placebo. No hypotheses will be tested in these subgroup analyses. See Section 7.0 for a list of tables presenting results by dose group.

#### 2.3 Missing Data Conventions

No missing value imputation will be used in this analysis. All analyses will be based on the observed data. For subjects that discontinue prior to Day 4 due to treatment related disability ("Rescue"), the observations collected at the time of rescue will be analyzed with the other Day 4 observations.

## 2.4 Interim Analyses

There are no interim analyses planned for this study.

## 2.5 Study Center Considerations in the Data Analysis

A study center is defined as a treatment administration site or group of treatment administration sites under the control and supervision of the same Principal Investigator (PI).

There will be no selective pooling of study centers in the analysis. All calculations will be made on the combined results of all centers.

#### 2.6 Documentation and Other Considerations

The data analyses will be conducted using SAS® Software, version 9.4 or later.

# 3.0 Analysis of Baseline Subject Characteristics

Baseline and demographic characteristics will be summarized by treatment and overall for all subjects in the safety population. Age and baseline weight will be displayed via summary statistics (mean, median, sample size, standard deviation, minimum, and maximum). Gender and ethnicity will be summarized via counts and percentages.

A detailed listing of demographics data for each subject will also be provided as shown in Appendix B.

# 4.0 Analysis of Efficacy

# 4.1 Description of Efficacy Variables

# 4.1.1 Primary Efficacy Variables

The co-primary efficacy variables for the study are the following:

- Subject Global Impression (SGI) score
- Quantitative Myasthenia Gravis (QMG) score

The calculations and analyses pertaining to each of the above variables are shown in Section 4.2.1.

#### 4.1.2 Secondary and Exploratory Efficacy Variables

The secondary and exploratory efficacy variables are the following:

- Clinical Global Impression of Improvement (CGI-I) score (secondary)
- Triple Timed Up and Go (3TUG) result (exploratory)
- Subject most bothersome symptom question (exploratory)
- QMG limb domains (exploratory)

The calculations and analyses pertaining to each of the above variables are shown in Section 4.2.2.

## 4.2 Analysis of Efficacy Variables

# 4.2.1 Primary Efficacy Analysis

Primary efficacy analyses will be conducted on the FAS and PP populations, with the FAS population serving as the primary analysis set. For both primary efficacy variables, change from baseline (CFB) will be computed as the post-treatment result (Day 4) minus the Baseline result (Day 0). The post-treatment result will be the result obtained on Day 4, unless the subject discontinued treatment early, in which case the post-treatment result may be obtained at an earlier time point.

Summary statistics for the QMG Day 0 assessment, QMG Day 4 assessment, and the corresponding CFB will be presented by treatment. The analysis of CFB for Total QMG Score is a co-primary efficacy endpoint and analysis will be performed by fitting a fixed effects linear model to the data with CFB as the response. The model will include terms for treatment and QMG at Baseline. The following test comparing the least squares (LS) means will be conducted to evaluate the treatment effect:

H<sub>A,0</sub>: LSMeanQMG(A) = LSMeanQMG(P) vs.
H<sub>A,1</sub>: LSMeanQMG(A) ≠ LSMeanQMG(P),

where LSMeanQMG(A) is the QMG LS mean of the amifampridine treatment group and LSMeanQMG(P) is the QMG LS mean of the placebo treatment group.

The raw individual QMG scores (each individual QMG domain) for Day 0, Day 4, and CFB will be summarized by treatment and dose within treatment. Additional between-treatment comparisons for several of the individual QMG domains, and the sum of these domains, will be performed using a fixed effects linear model as an exploratory endpoint. No inferential procedures will be performed on the other QMG domains. See section 4.2.2 for details.

Summary statistics for SGI score and the corresponding CFB will be presented by treatment. The analysis of CFB for SGI is a co-primary efficacy endpoint and analysis will be performed by fitting a fixed effects linear model to the data with CFB as the response. The model will include terms for treatment and SGI at Baseline. The following test comparing the LS means will be conducted to evaluate the treatment effect:

 $H_{B,0}$ : LSMeanSGI(A) = LSMeanSGI(P) vs.  $H_{B,1}$ : LSMeanSGI(A)  $\neq$  LSMeanSGI(P),

where LSMeanSGI(A) is the SGI LS mean of the amifampridine treatment group and LSMeanSGI(P) is the SGI LS mean of the placebo treatment group.

A sensitivity analysis of the co-primary endpoints will be conducted to evaluate the patterns of early treatment discontinuation. For each co-primary endpoint, a randomization test will be conducted to determine if the results from the primary analysis are supported. The randomization test is an alternative to a full permutation, and will evaluate the fixed effects model specified above using permutations of the treatment group assignments. If early discontinuations are not associated with treatment, then it is expected that the p-value resulting from the randomization test will yield the same statistical interpretation as the p-value resulting from the primary analysis.

A data listing of the primary efficacy data will be constructed as shown in Appendix B.

# 4.2.2 Secondary and Exploratory Efficacy Analyses

Secondary and exploratory efficacy analyses will be conducted on the FAS and PP populations, with the FAS population serving as the primary analysis set.

#### Clinical Global Impression of Improvement (CGI-I)

CGI-I scores will be summarized by treatment group using descriptive statistics. A Wilcoxon Rank Sum Test will be conducted to assess for treatment group differences.

## Triple Timed Up and Go (3TUG)

The number and proportion of subjects with at least a 20% increase in average time for 3TUG (i.e., a success) at Day 4 relative to Day 0 will be presented by treatment. For those subjects that are unable to complete the Day 4 assessment due to disability related to their disease, a success will be assigned to the subject by the site at the time of testing. The proportion will be computed in two ways: 1) using all subjects in the analysis population with Day 0 data as the denominator, regardless of whether or not they completed the Day 4 assessment; and 2) using only those subjects in the analysis population who completed both the Day 0 and Day 4 assessments. For each approach in calculating the proportion, a two-sided Fisher's Exact Test will be conducted to

test for a significant difference in the success proportions between treatment groups.

# **Patient Most Bothersome Symptom Question**

For the Patient Most Bothersome Symptom (PMBS) question, change from baseline (CFB) will be computed as the post-treatment response (Day 4) minus the Baseline response (Day 0). The post-treatment response will be the result obtained on Day 4, unless the subject discontinued treatment early, in which case the post-treatment response may be obtained at an earlier time point.

Summary statistics for the PMBS Day 0 response, PBMS Day 4 response, and the corresponding CFB will be presented by treatment. The analysis of CFB for PMBS Score will be performed using Wilcoxon's Rank Sum Test.

#### **QMG Limb Domains**

Descriptive statistics for Day 0, Day 4, and CFB for the sum of the QMG scores for Right arm outstretched, Left arm outstretched, Right leg outstretched, and Left leg outstretched will be presented by treatment. As was described in section 4.2.1, summary statistics will be presented for each of these for individual domains. The CFB for each of these four individual domains, and for the sum of these four domains, will be performed by fitting a fixed effects linear model to the data with CFB as the response. The model will include terms for treatment and QMG score of the respective individual domain, or sum of these four domains, as applicable, at Baseline. The following test comparing the least squares (LS) means will be conducted to evaluate the treatment effect:

H<sub>C,0</sub>: LSMeanQMG(A) = LSMeanQMG(P) vs.
H<sub>C,1</sub>: LSMeanQMG(A) ≠ LSMeanQMG(P),

where LSMeanQMG(A) is the QMG LS mean of the amifampridine treatment group and LSMeanQMG(P) is the QMG LS mean of the placebo treatment group for each individual QMG domain described above, or sum of these 4 domains. A sensitivity analysis by a randomization test for the QMG limb domain analyses is not required.

All secondary and exploratory efficacy data will be listed as shown in Appendix B.

# 5.0 Analysis of Safety

The safety variables for this study are:

- Adverse events (AE)
- Vital signs (screening, Days 1-4)

- Physical examination (at screening only)
- Concomitant medications

#### **Adverse Events**

All AEs will be observed for each subject from enrollment until termination from the study. Prior to analysis, all AEs will be coded using MedDRA. Based on these coded terms, treatment emergent AEs (TEAEs) will be summarized using system organ class and preferred term by treatment and overall for all subjects in the safety population. This analysis will be repeated for serious TEAEs (TESAEs).

TEAEs will also be summarized by severity and relationship to IP. An overall summary table will provide the highest relationship and maximum severity observed per subject, as well as the counts of subjects with at least one TESAE.

All AEs will be listed, regardless of whether or not they were treatment emergent. AEs having an end date prior to signing the informed consent for this study will not be displayed in the AE data listings.

# **Vital Signs**

Summary statistics (mean, median, sample size, standard deviation, minimum, and maximum) will be computed on the raw and change from baseline values for each vital sign parameter by time point, for each treatment. The screening time point will serve as baseline. If there are multiple vital signs taken at any time point, then the latest set of vital signs will be used for the analysis. All vital sign data will be listed.

#### Physical Exam

The physical exam data collected at screening will be listed.

#### **Concomitant Medications**

A table of the WHO-coded medications will be constructed by treatment group and overall with medications summarized by level 3 anatomical therapeutic chemical (ATC) term and Preferred Term . The number and percent of subjects on each drug will be summarized. A data listing for all concomitant medications will be provided.

# 6.0 Other Relevant Data Analyses/Summaries

# **6.1 Subject Completion**

A table will be constructed with counts of screen failures and enrolled subjects. Of those enrolled, counts and percentages of the number of subjects withdrawing from the study before study completion and the number completing the study will be displayed. For those subjects that withdraw before completion of the study, counts and percentages of the reasons for withdrawal will be tabulated. The

table will include summary counts and percentages by treatment. A data listing of all subject completion and withdrawal data will also be constructed.

# 6.2 Study Drug Administration and Compliance

Duration of treatment administration will be computed per subject as:

Duration (in days) = (Date of last dose) – (Date of first dose) + 1

Duration will be summarized using descriptive statistics by treatment group.

Compliance will be computed per subject as:

Compliance = 100%\*(Number consumed)/(Number prescribed),

where number prescribed is defined as the duration times the number of tablets to have been taken daily. Compliance will be summarized using descriptive statistics by treatment group.

#### 6.3 Patient Data Profiles

A Patient Data Profile listing will be provided. It will contain demographic information, randomization information, all endpoint assessments and laboratory measurements. See\_Appendix B, Data Listing 17 for full details. Some variation in the appearance of this table is acceptable to accommodate unformatted SAS® output provided that all information is present.

# 7.0 List of Analysis Tables, Figures and Listings

| Table<br>No. | Table Title | Included<br>in Final<br>Tables | Shown in<br>Appendix<br>B |
|---|---|---|---|
| 1 | Subject Disposition | X | X |
| 2 | Demographics and Baseline Data Summary Statistics – Continuous Variables (Safety Population) | Х | Х |
| 3 | Demographics and Baseline Data Summary Statistics – Categorical Variables (Safety Population) | Х | Х |
| 4 | Summary of Study Drug Administration and Compliance (Safety Population) | Х | Х |
| 5 | QMG Total Score Summary Statistics by Time Point (FAS Population) | Х | Х |
| 6 | QMG Total Score Summary Statistics by Time Point (PP Population) | Х | |
| 7 | QMG Total Score Summary Statistics by Time Point and Dose Group (FAS Population) | Х | Х |
| 8 | QMG Total Score Summary Statistics by Time Point and Dose Group (PP Population) | Х | |
| 9 | QMG Item Scores Summary Statistics by Time Point (FAS Population) | Х | х |
| 10 | QMG Item Scores Summary Statistics by Time Point (PP Population) | Х | |
| 11 | QMG Item Scores Summary Statistics by Time Point and Dose Group (FAS Population) | Х | Х |
| 12 | QMG Item Scores Summary Statistics by Time Point and Dose Group (PP Population) | Х | |
| 13 | QMG Total Score CFB Analysis (FAS Population) | Х | Х |
| 14 | QMG Total Score CFB Analysis (PP Population) | Х | |
| 15 | QMG Item Scores CFB Analysis (FAS Population) | Х | Х |
| 16 | QMG Item Scores CFB Analysis (PP Population) | Х | |
| 17 | SGI Score Summary Statistics by Time Point (FAS Population) | Х | Х |
| 18 | SGI Score Summary Statistics by Time Point (PP Population) | Х | |
| 19 | SGI Score Summary Statistics by Time Point and Dose Group (FAS Population) | Х | х |
| 20 | SGI Score Summary Statistics by Time Point and Dose Group (PP Population) | Х | |
| 21 | SGI Score CFB (FAS Population) | Х | Х |
| 22 | SGI Score CFB Analysis (PP Population) | Х | |
| 23 | QMG Total Score and SGI Score Sensitivity Analysis (FAS Population) | Х | х |
| 24 | QMG Total Score and SGI Score Sensitivity Analysis (PP Population) | Х | |
| 25 | CGI-I Scores Summary Statistics (FAS Population) | Х | Х |
| 26 | CGI-I Scores Summary Statistics (PP Population) | Х | |
| 27 | CGI-I Scores Summary Statistics by Dose Group (FAS Population) | Х | Х |
| 28 | CGI-I Scores Summary Statistics by Dose Group (PP Population) | Х | |

| Table<br>No. | Table Title | Included in Final Tables | Shown in<br>Appendix<br>B |
|---|---|---|---|
| 29 | Number and Proportion of Subjects with ≥ 20% Increase in 3TUG Average Time (FAS Population) | Х | Х |
| 30 | Number and Proportion of Subjects with ≥ 20% Increase in 3TUG Average Time (PP Population) | Х | |
| 31 | Number and Proportion of Subjects with ≥ 20% Increase in 3TUG Average Time by Dose Group (FAS Population) | × | X |
| 32 | Number and Proportion of Subjects with ≥ 20% Increase in 3TUG Average Time by Dose Group (PP Population) | × | |
| 33 | Summary of Patient Most Bothersome Symptom (FAS Population) | × | х |
| 34 | Summary of Patient Most Bothersome Symptom (PP Population) | Х | |
| 35 | Summary of Patient Most Bothersome Symptom by Dose Group (FAS Population) | Х | Х |
| 36 | Summary of Patient Most Bothersome Symptom by Dose Group (PP Population) | Х | |
| 37 | QMG Total Score Summary Statistics by Limb Domain and Time Point (FAS Population) | Х | Х |
| 38 | QMG Total Score Summary Statistics by Limb Domain and Time Point (PP Population) | Х | |
| 39 | Limb Domain Specific QMG Total Score CFB Analysis (FAS Population) | Х | Х |
| 40 | Limb Domain Specific QMG Total Score CFB Analysis (PP Population) | Х | |
| 41 | Number and Percent of Subjects with Treatment<br>Emergent Adverse Events (Safety Population) | Х | Х |
| 42 | Number and Percent of Subjects with Treatment<br>Emergent Adverse Events by Dose Level (Safety<br>Population) | Х | х |
| 43 | Summary of Treatment Emergent Adverse Events (Safety Population) | Х | Х |
| 44 | Number and Percent of Subjects with Serious Treatment<br>Emergent Adverse Events (Safety Population) | Х | Х |
| 45 | Number and Percent of Subjects with Treatment Emergent Adverse Events by Relationship to Treatment (Safety Population) | Х | Х |
| 46 | Number and Percent of Subjects with Treatment Emergent Adverse Events by Severity Grade (Safety Population) | Х | Х |
| 47 | Vital Sign Parameters Summary Statistics (Safety Population) | Х | Х |
| 48 | Number and Percent of Subjects Taking Concomitant Medications by ATC Level 3 and Preferred Term (Safety Population) | Х | Х |

| Listing<br>No. | Data Listing Title | Included<br>in Final<br>Listings | Shown in<br>Appendix B |
|---|---|---|---|
| DL1 | Subject Disposition Data Listing | X | X |
| DL2 | Protocol Deviations Data Listing | X | X |
| DL3 | Demographics Data Listing | X | X |
| DL4 | Subjects Excluded from FAS Population Data Listing | Х | Х |
| DL5 | Subjects Excluded from PP Population Data Listing | Х | Х |
| DL6 | Medical History Data Listing | Х | X |
| DL7 | Prior and Concomitant Medications Data Listing | Х | X |
| DL8 | Adverse Events Data Listing | Х | X |
| DL9 | Physical Exam Data Listing | Х | X |
| DL10 | Vital Signs Data Listing | Х | X |
| DL11 | Study Drug Administration Data Listing | Х | X |
| DL12 | SGI Data Listing | Х | X |
| DL13 | QMG Data Listing | Х | X |
| DL14 | CGI-I Data Listing | Х | X |
| DL15 | 3TUG Data Listing | Х | X |
| DL16 | Patient Most Bothersome Symptom Data Listing | Х | X |
| DL17 | Patient Data Profile | Х | X |

# 8.0 References

Cassell, David. A Randomization-test Wrapper for SAS® PROCs. Paper 251-27, (2002) SUGI 27 Proceedings.

http://www2.sas.com/proceedings/sugi27/p251-27.pdf, doi:2017-06-22.

# Appendix A – Tables, Figures and Listing Specifications

#### Orientation

Tables, figures, and listings will be displayed in landscape.

## Margins

Margins will be 1 inch on all sides. Table, figure, and listing boundaries will not extend into the margins.

#### **Font**

Courier New, 8 point.

#### **Headers**

The table number will be on the second line of the title area. The title area will contain the Sponsor name, the study number, and the name of the table. The title area will contain the page number (Page x of y) on the far right, one line above the name of the table.

#### **Footers**

- The first line will be a solid line.
- Next will be any footnotes regarding information displayed in the table.
- The last line will display the name of the SAS program that generated the table and (if applicable) the source data reference.

#### **Table Disclaimer**

The format of the mock tables shown in the appendix of this Statistical Analysis Plan (SAP) will be the format of the deliverable tables to the extent that Word document constructed tables can match production tables produced by SAS. This formatting includes the content and format of the header and footer areas of the tables. The Sponsor agrees to the format of the tables as shown in the appendix.

Further programming charges will be applicable for changes in the format of tables (including title statements, notes, data dependent footnotes, etc.) made after the approval of the SAP.

# **Missing Values**

All missing values will be displayed on the output tables/listings as blanks.

# **Computation Values for Study Dates**

The date format to be used is dd-mmm-yyyy. Missing parts of dates are not shown (e.g., for a missing day value, the value displayed is in mmm-yyyy format). When date computations are necessary, the following table indicates the substitutions used in order to make those computations.

| Scenario | Value Used for Computations |
|---|---|
| Start date – Missing month and day values | January 1 of the indicated year |
| Start date – Missing day values | The first day of the indicated month |
| Stop date – Missing month and day values | December 31 of the indicated year |
| Stop date – Missing day values | The last day of the indicated month |

# Appendix B – Table Shells

Page x of y

Table 1. Subject Disposition
Catalyst Pharmaceuticals, Inc. - LMS-003

| | | Amifampridine | Placebo | Overall |
|---|---|---|---|---|
| Screen Failures | | | | XX |
| Enrolled | | XX | xx | xx |
| | Low Dose (< 60 mg/day) | xx (xxx%) | xx (xxx%) | xx (xxx%) |
| | High Dose ( $\geq$ 60 mg/day) | xx (xxx%) | xx (xxx%) | xx (xxx%) |
| Completed | | xx (xxx%) | xx (xxx%) | xx (xxx%) |
| | Low Dose (< 60 mg/day) | xx (xxx%) | xx (xxx%) | xx (xxx%) |
| | High Dose ( $\geq$ 60 mg/day) | xx (xxx%) | xx (xxx%) | xx (xxx%) |
| ithdrawn | | xx (xxx%) | xx (xxx%) | xx (xxx%) |
| | Low Dose (< 60 mg/day) | xx (xxx%) | xx (xxx%) | xx (xxx%) |
| | High Dose ( $\geq$ 60 mg/day) | xx (xxx%) | xx (xxx%) | xx (xxx%) |
| eason for Withdrawal | Adverse Event | xx (xxx%) | xx (xxx%) | xx (xxx%) |
| | Low Dose (< 60 mg/day) | xx (xxx%) | xx (xxx%) | xx (xxx%) |
| | High Dose ( $\geq$ 60 mg/day) | xx (xxx%) | xx (xxx%) | xx (xxx%) |
| | Lost To Follow-Up | xx (xxx%) | xx (xxx%) | xx (xxx%) |
| | Low Dose (< 60 mg/day) | xx (xxx%) | xx (xxx%) | xx (xxx%) |
| | High Dose (≥ 60 mg/day) | xx (xxx%) | xx (xxx%) | xx (xxx%) |
| | Death | xx (xxx%) | xx (xxx%) | xx (xxx% |
| | Low Dose (< 60 mg/day) | xx (xxx%) | xx (xxx%) | xx (xxx% |
| | High Dose (≥ 60 mg/day) | xx (xxx%) | xx (xxx%) | xx (xxx%) |
| | Physician Decision | xx (xxx%) | xx (xxx%) | xx (xxx%) |
| | Low Dose (< 60 mg/day) | xx (xxx%) | xx (xxx%) | xx (xxx%) |
| | High Dose ( <u>&gt;</u> 60 mg/day) | xx (xxx%) | xx (xxx%) | xx (xxx%) |
| | Protocol Deviation | xx (xxx%) | xx (xxx%) | xx (xxx%) |
| | Low Dose (< 60 mg/day) | xx (xxx%) | xx (xxx%) | xx (xxx%) |
| | High Dose (≥ 60 mg/day) | xx (xxx%) | xx (xxx%) | xx (xxx%) |
| | Study Terminated by Sponsor | xx (xxx%) | xx (xxx%) | xx (xxx%) |
| | Low Dose (< 60 mg/day) | xx (xxx%) | xx (xxx%) | xx (xxx%) |
| | High Dose ( $\geq$ 60 mg/day) | xx (xxx%) | xx (xxx%) | xx (xxx%) |
| | Withdrawal by Subject | xx (xxx%) | xx (xxx%) | xx (xxx%) |
| | Low Dose (< 60 mg/day) | xx (xxx%) | xx (xxx%) | xx (xxx%) |
| | High Dose ( $\geq$ 60 mg/day) | xx (xxx%) | xx (xxx%) | xx (xxx%) |
| | Other | xx (xxx%) | xx (xxx%) | xx (xxx%) |
| | Low Dose (< 60 mg/day) | xx (xxx%) | xx (xxx%) | xx (xxx%) |
| | High Dose (> 60 mg/day) | xx (xxx%) | xx (xxx%) | xx (xxx%) |

The denominator for all percentages in the table is the number of enrolled subjects in the pertinent treatment/dose group and overall.

Table Creation Date: (DD-MMM-YYYY)
Source Program: xxxxxxx.sas
Source Listing: Data Listing 1

Page x of y

Table 2. Demographics and Baseline Data Summary Statistics - Continuous Variables Catalyst Pharmaceuticals, Inc. - LMS-003 Safety Population (N=xxx)

| Variable | Treatment Group | Mean | Std Dev | n | Min | Max | Median |
|---|---|---|---|---|---|---|---|
| Age (years) | Amifampridine | XXX | XXX | XXX | XXX | XXX | XXX |
| | Low Dose (< 60 mg/day) | XXX | XXX | XXX | XXX | XXX | XXX |
| | High Dose ( <u>&gt;</u> 60 mg/day) | XXX | XXX | XXX | XXX | XXX | XXX |
| | Placebo | XXX | XXX | XXX | XXX | XXX | XXX |
| | Low Dose (< 60 mg/day) | XXX | XXX | XXX | XXX | XXX | XXX |
| | High Dose (> 60 mg/day) | XXX | XXX | XXX | XXX | XXX | XXX |
| | Overall | XXX | XXX | XXX | XXX | XXX | xxx |
| Baseline Weight (kg) | Amifampridine | xxx | xxx | xxx | xxx | xxx | xxx |
| | Low Dose (< 60 mg/day) | XXX | XXX | XXX | XXX | XXX | XXX |
| | High Dose (> 60 mg/day) | XXX | XXX | XXX | XXX | XXX | XXX |
| | Placebo | XXX | XXX | XXX | XXX | XXX | XXX |
| | Low Dose (< 60 mg/day) | XXX | XXX | XXX | XXX | XXX | XXX |
| | High Dose (> 60 mg/day) | XXX | XXX | XXX | XXX | XXX | XXX |
| | Overall | XXX | XXX | XXX | XXX | XXX | XXX |

Table Creation Date: (DD-MMM-YYYY)

Source Program: xxxxxxx.sas Source Listing: Data Listing 3

Page x of y

Table 3. Demographics and Baseline Data Summary Statistics - Categorical Variables Catalyst Pharmaceuticals, Inc. - LMS-003 Safety Population (N=xxx)

| Demographics<br>Variable | Category | Amifampridine (N=xxx) | Placebo<br>(N=xxx) | Overall (N=xxx) |
|---|---|---|---|---|
| - | <u> </u> | , | · | |
| Gender | Male | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |
| | Low Dose (< 60 mg/day) | xx (xxx%a) | xx (xxx%) | xx (xxx%) |
| | High Dose (> 60 mg/day) | xx (xxx%) | xx (xxx%) | xx (xxx%) |
| | Female | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |
| | Low Dose (< 60 mg/day) | xx (xxx%) | xx (xxx%) | xx (xxx%) |
| | High Dose ( <u>&gt;</u> 60 mg/day) | xx (xxx%) | xx (xxx%) | xx (xxx%) |
| Ethnicity | Hispanic or Latino | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |
| | Low Dose (< 60 mg/day) | xx (xxx%) | xx (xxx%) | xx (xxx%) |
| | High Dose (> 60 mg/day) | xx (xxx%) | xx (xxx%) | xx (xxx%) |
| | Not Hispanic or Latino | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |
| | Low Dose (< 60 mg/day) | xx (xxx%) | xx (xxx%) | xx (xxx%) |
| | High Dose (> 60 mg/day) | xx (xxx%) | xx (xxx%) | xx (xxx%) |

Table Creation Date: (DD-MMM-YYYY)
Source Program: xxxxxxx.sas

Source Listing: Data Listing 3

<sup>&</sup>lt;sup>a</sup> Denominator for treatment/class/dose percentages is the treatment/class/dose level total.

Page x of y

Table 4. Summary of Study Drug Administration and Compliance Catalyst Pharmaceuticals, Inc. - LMS-003 Safety Population (N=xxx)

| | | Amifampridine | Placebo |
|-----------------|------------------|---------------|-----------|
| | Statistic | (N=xxx) | (N=xxx) |
| Duration (days) | n | XXX | XXX |
| | Mean (SD) | xxx (xxx) | xxx (xxx) |
| | Median | XXX | XXX |
| | Minimum, Maximum | xxx, xxx | XXX, XXX |
| Compliance (%) | n | xxx | xxx |
| | Mean (SD) | xxx (xxx) | xxx (xxx) |
| | Median | xxx | XXX |
| | Minimum, Maximum | xxx, xxx | xxx, xxx |

Table Creation Date: (DD-MMM-YYYY)

Source Program: xxxxxxx.sas Source Listing: Data Listing 11

Page x of y

Table 5. QMG Total Score Summary Statistics by Time Point Catalyst Pharmaceuticals, Inc. - LMS-003 FAS Population (N=xxx)

| | | | | Std | | | | |
|---|---|---|---|---|---|---|---|---|
| Treatment | Time Point <sup>a</sup> | Data Type <sup>b</sup> | Mean | Dev | n | Min | Max | Median |
| Amifampridine | Day 0 (Baseline) | RAW | xxx | xxx | xxx | xxx | xxx | XXX |
| - | Post-Baseline | RAW | XXX | XXX | XXX | XXX | XXX | XXX |
| | | CFB | XXX | XXX | XXX | XXX | XXX | XXX |
| Placebo | Day 0 (Baseline) | RAW | xxx | xxx | xxx | xxx | xxx | xxx |
| | Post-Baseline | RAW | XXX | XXX | XXX | XXX | XXX | XXX |
| | | CFB | XXX | XXX | xxx | XXX | XXX | XXX |

Table Creation Date: (DD-MMM-YYYY)
Source Program: xxxxxxx.sas

Source Listing: Data Listing 14

<sup>&</sup>lt;sup>a</sup> The post-treatment result will be the result obtained on Day 4, unless the subject discontinued treatment early, in which case the post-treatment result may be obtained at an earlier time point.

 $<sup>^{\</sup>mathrm{b}}$  RAW = observed data entered in the database; CFB = change from baseline.

Page x of y

Table 7. QMG Total Score Summary Statistics by Time Point and Dose Group Catalyst Pharmaceuticals, Inc. - LMS-003 FAS Population (N=xxx)

| | | | Data | | Std | | | | |
|---|---|---|---|---|---|---|---|---|---|
| Treatment | Dose Group | Time Point <sup>a</sup> | Type <sup>b</sup> | Mean | Dev | n | Min | Max | Median |
| Amifampridine | | | | | | | | | |
| | Low Dose (< 60mg/day) | Day 0 (Baseline) | RAW | XXX | XXX | XXX | XXX | XXX | XXX |
| | | Post-Baseline | RAW | XXX | XXX | XXX | XXX | XXX | XXX |
| | | | CFB | XXX | XXX | XXX | XXX | XXX | XXX |
| | High Dose ( $\geq$ 60mg/day) | Day 0 (Baseline) | RAW | XXX | XXX | XXX | XXX | XXX | XXX |
| | | Post-Baseline | RAW | XXX | XXX | XXX | XXX | XXX | XXX |
| | | | CFB | XXX | XXX | XXX | XXX | XXX | XXX |
| | All Doses | Day 0 (Baseline) | RAW | XXX | XXX | XXX | XXX | XXX | XXX |
| | | Post-Baseline | RAW | XXX | XXX | XXX | XXX | XXX | XXX |
| | | | CFB | XXX | XXX | XXX | XXX | XXX | XXX |
| Placebo | | | | | | | | | |
| | Low Dose (< 60mg/day) | Day 0 (Baseline) | RAW | XXX | XXX | XXX | XXX | XXX | XXX |
| | | Post-Baseline | RAW | XXX | XXX | XXX | XXX | XXX | XXX |
| | | | CFB | XXX | XXX | XXX | XXX | XXX | XXX |
| | High Dose ( $\geq$ 60mg/day) | Day 0 (Baseline) | RAW | XXX | XXX | XXX | XXX | XXX | XXX |
| | | Post-Baseline | RAW | XXX | XXX | XXX | XXX | XXX | XXX |
| | | | CFB | XXX | XXX | XXX | XXX | XXX | XXX |
| | All Doses | Day 0 (Baseline) | RAW | XXX | XXX | XXX | XXX | XXX | XXX |
| | | Post-Baseline | RAW | XXX | XXX | XXX | XXX | XXX | XXX |
| | | | CFB | XXX | XXX | XXX | XXX | XXX | XXX |

Table Creation Date: (DD-MMM-YYYY)

Source Program: xxxxxxx.sas Source Listing: Data Listing 14

<sup>&</sup>lt;sup>a</sup> The post-treatment result will be the result obtained on Day 4, unless the subject discontinued treatment early, in which case the post-treatment result may be obtained at an earlier time point.

 $<sup>^{\</sup>mathrm{b}}$  RAW = observed data entered in the database; CFB = change from baseline.

Page x of y

Table 9. QMG Item Scores Summary Statistics by Time Point Catalyst Pharmaceuticals, Inc. - LMS-003 FAS Population (N=xxx)

| | | | | | Std | | | | |
|---|---|---|---|---|---|---|---|---|---|
| Treatment | QMG Item <sup>a</sup> | Time Point <sup>b</sup> | Data Type <sup>b</sup> | Mean | Dev | n | Min | Max | Median |
| Amifampridine | xxxxxxxxx | Day 0 (Baseline) | RAW | xxx | xxx | xxx | xxx | xxx | xxx |
| IIMII I I I I I I I I I I I I I I I I I | *************************************** | Post-Baseline | RAW | XXX | XXX | XXX | XXX | XXX | XXX |
| | | | CFB | XXX | XXX | XXX | XXX | XXX | XXX |
| Placebo | xxxxxxxxx | Day 0 (Baseline) | RAW | XXX | xxx | xxx | xxx | xxx | XXX |
| | | Post-Baseline | RAW | XXX | XXX | XXX | XXX | XXX | xxx |
| | | | CFB | XXX | XXX | XXX | XXX | XXX | XXX |

Table Creation Date: (DD-MMM-YYYY)
Source Program: xxxxxxx.sas

Source Listing: Data Listing 14

<sup>&</sup>lt;sup>a</sup> Table excludes limb domain items which are summarized on separate tables.

<sup>&</sup>lt;sup>b</sup> The post-treatment result will be the result obtained on Day 4, unless the subject discontinued treatment early, in which case the post-treatment result may be obtained at an earlier time point.

b RAW = observed data entered in the database; CFB = change from baseline.

Page x of y

Table 11. QMG Item Scores Summary Statistics by Time Point and Dose Group Catalyst Pharmaceuticals, Inc. - LMS-003 FAS Population (N=xxx)

QMG Parameter = xxxxxxxxxxxx

C+ 4

| | | | | | Std | | | | |
|---|---|---|---|---|---|---|---|---|---|
| Treatment | Dose Group | Time Point <sup>a</sup> | Data Type <sup>b</sup> | Mean | Dev | n | Min | Max | Median |
| Amifampridine | | | | | | | | | |
| | Low Dose (< 60mg/day) | Day 0 (Baseline) | RAW | XXX | XXX | XXX | XXX | XXX | XXX |
| | | Post-Baseline | RAW | XXX | XXX | XXX | XXX | XXX | XXX |
| | | | CFB | XXX | XXX | XXX | XXX | XXX | XXX |
| | High Dose (> 60mg/day) | Day 0 (Baseline) | RAW | XXX | XXX | XXX | XXX | XXX | XXX |
| | | Post-Baseline | RAW | XXX | XXX | XXX | XXX | XXX | XXX |
| | | | CFB | XXX | XXX | XXX | XXX | XXX | XXX |
| | All Doses | Day 0 (Baseline) | RAW | XXX | XXX | XXX | XXX | XXX | XXX |
| | | Post-Baseline | RAW | XXX | XXX | XXX | XXX | XXX | XXX |
| | | | CFB | XXX | XXX | XXX | XXX | XXX | XXX |
| Placebo | | | | | | | | | |
| | Low Dose (< 60mg/day) | Day 0 (Baseline) | RAW | XXX | XXX | XXX | XXX | XXX | XXX |
| | | Post-Baseline | RAW | XXX | XXX | XXX | XXX | XXX | XXX |
| | | | CFB | XXX | XXX | XXX | XXX | XXX | XXX |
| | High Dose (> 60mg/day) | Day 0 (Baseline) | RAW | XXX | XXX | XXX | XXX | XXX | XXX |
| | | Post-Baseline | RAW | XXX | XXX | XXX | XXX | XXX | XXX |
| | | | CFB | XXX | XXX | XXX | XXX | XXX | XXX |
| | All Doses | Day 0 (Baseline) | RAW | XXX | XXX | XXX | XXX | XXX | XXX |
| | | Post-Baseline | RAW | XXX | XXX | XXX | XXX | XXX | XXX |
| | | | CFB | XXX | XXX | XXX | XXX | XXX | XXX |

# **Table repeats per QMG Parameter**

Table Creation Date: (DD-MMM-YYYY)

Source Program: xxxxxxx.sas Source Listing: Data Listing 14

<sup>&</sup>lt;sup>a</sup> The post-treatment result will be the result obtained on Day 4, unless the subject discontinued treatment early, in which case the post-treatment result may be obtained at an earlier time point.

b RAW = observed data entered in the database; CFB = change from baseline.

Page x of y

#### Table 13. QMG Total Score CFB Analysis Catalyst Pharmaceuticals, Inc. - LMS-003 FAS Population (N=xxx)

| Statistic <sup>a</sup> | Amifampridine | Placebo |
|---|---|---|
| n | xxx | xxx |
| Least Squares (LS) Mean of Change from Baseline (CFB) | xxx | xxx |
| Between-Treatment Difference in LS Means | xxx | |
| 95% CI for Between-Treatment Difference in LS Means | (xxx, xxx) | |
| P-value for Between-Treatment Difference in LS Means | XXX | |

<sup>a</sup> CFB for QMG total score was modeled as the response, with fixed effects terms for treatment and QMG at Baseline. Table Creation Date: (DD-MMM-YYYY)

xxxxxxx.sas

Source Listing: Data Listing 14

Page x of y

#### Table 15. QMG Item Scores CFB Analysis Catalyst Pharmaceuticals, Inc. - LMS-003 FAS Population (N=xxx)

| QMG Item | Statistic <sup>a</sup> | Amifampridine | Placebo |
|---|---|---|---|
| xxxxxxxx | n | xxx | xxx |
| | Least Squares (LS) Mean of Change from Baseline (CFB) | XXX | xxx |
| | Between-Treatment Difference in LS Means | xxx | |
| | 95% CI for Between-Treatment Difference in LS Means | (xxx, xxx) | |
| | P-value for Between-Treatment Difference in LS Means | XXX | |

Table Creation Date: (DD-MMM-YYYY) Source Program: xxxxxxx.sas Source Listing: Data Listing 14

 $<sup>\</sup>overline{a}$  CFB for QMG item score was modeled as the response, with fixed effects terms for treatment and QMG at Baseline. A separate model was run for each QMG item.

Page x of y

# Table 17. SGI Score Summary Statistics by Time Point Catalyst Pharmaceuticals, Inc. - LMS-003 FAS Population (N=xxx)

| | | | | Std | | | | |
|---|---|---|---|---|---|---|---|---|
| Treatment | Time Point <sup>a</sup> | Data Type <sup>b</sup> | Mean | Dev | n | Min | Max | Median |
| - 15 131 | - 0 (- 1) | | | | | | | |
| Amifampridine | Day O (Baseline) | RAW | XXX | XXX | XXX | XXX | XXX | XXX |
| | Post-Baseline | RAW | XXX | XXX | XXX | XXX | XXX | XXX |
| | | CFB | XXX | XXX | XXX | XXX | XXX | XXX |
| Placebo | Day 0 (Baseline) | RAW | xxx | xxx | xxx | XXX | xxx | xxx |
| | Post-Baseline | RAW | XXX | XXX | XXX | XXX | XXX | XXX |
| | | CFB | XXX | XXX | XXX | XXX | XXX | XXX |

Table Creation Date: (DD-MMM-YYYY)
Source Program: xxxxxxx.sas

Source Program: xxxxxxx.sas Source Listing: Data Listing 13

<sup>&</sup>lt;sup>a</sup> The post-treatment result will be the result obtained on Day 4, unless the subject discontinued treatment early, in which case the post-treatment result may be obtained at an earlier time point.

b RAW = observed data entered in the database; CFB = change from baseline.

Page x of y

Table 19. SGI Score Summary Statistics by Time Point and Dose Group Catalyst Pharmaceuticals, Inc. - LMS-003

FAS Population (N=xxx)

| | | | | | Std | | | | |
|---|---|---|---|---|---|---|---|---|---|
| Treatment | Dose Group | Time Point <sup>a</sup> | Data Type <sup>b</sup> | Mean | Dev | n | Min | Max | Median |
| Amifampridine | | | | | | | | | |
| | Low Dose (< 60mg/day) | Day 0 (Baseline) | RAW | XXX | XXX | XXX | XXX | XXX | XXX |
| | | Post-Baseline | RAW | XXX | XXX | XXX | XXX | XXX | XXX |
| | | | CFB | XXX | XXX | XXX | XXX | XXX | XXX |
| | High Dose (> 60mg/day) | Day 0 (Baseline) | RAW | XXX | XXX | XXX | XXX | XXX | XXX |
| | | Post-Baseline | RAW | XXX | XXX | XXX | XXX | XXX | XXX |
| | | | CFB | XXX | XXX | XXX | XXX | XXX | XXX |
| | All Doses | Day 0 (Baseline) | RAW | XXX | XXX | XXX | XXX | XXX | XXX |
| | | Post-Baseline | RAW | XXX | XXX | XXX | XXX | XXX | XXX |
| | | | CFB | XXX | XXX | XXX | XXX | XXX | XXX |
| Placebo | | | | | | | | | |
| | Low Dose (< 60mg/day) | Day 0 (Baseline) | RAW | XXX | XXX | XXX | XXX | XXX | XXX |
| | | Post-Baseline | RAW | XXX | XXX | XXX | XXX | XXX | XXX |
| | | | CFB | XXX | XXX | XXX | XXX | XXX | XXX |
| | High Dose (> 60mg/day) | Day 0 (Baseline) | RAW | XXX | XXX | XXX | XXX | XXX | XXX |
| | | Post-Baseline | RAW | XXX | XXX | XXX | XXX | XXX | XXX |
| | | | CFB | XXX | XXX | XXX | XXX | XXX | XXX |
| | All Doses | Day 0 (Baseline) | RAW | XXX | XXX | XXX | XXX | XXX | XXX |
| | | Post-Baseline | RAW | XXX | XXX | XXX | XXX | XXX | XXX |
| | | | CFB | XXX | XXX | XXX | XXX | XXX | XXX |

Table Creation Date: (DD-MMM-YYYY)
Source Program: xxxxxxx.sas

Source Program: xxxxxxx.sas Source Listing: Data Listing 13

<sup>&</sup>lt;sup>a</sup> The post-treatment result will be the result obtained on Day 4, unless the subject discontinued treatment early, in which case the post-treatment result may be obtained at an earlier time point.

b RAW = observed data entered in the database; CFB = change from baseline.

Page x of y

# Table 21. SGI Score CFB Analysis Catalyst Pharmaceuticals, Inc. - LMS-003 FAS Population (N=xxx)

| Statistic <sup>a</sup> | Amifampridine | Placebo |
|---|---|---|
| n | xxx | xxx |
| Least Squares (LS) Mean of Change from Baseline (CFB) | xxx | xxx |
| Between-Treatment Difference in LS Means | xxx | |
| 95% CI for Between-Treatment Difference in LS Means | (xxx, xxx) | |
| P-value for Between-Treatment Difference in LS Means | XXX | |

<sup>a</sup> CFB for SGI score was modeled as the response, with fixed effects terms for treatment and QMG at Baseline.

Table Creation Date: (DD-MMM-YYYY)
Source Program: xxxxxxx.sas

Source Program: xxxxxxx.sas Source Listing: Data Listing 13

Page x of y

Table 23. QMG Total Score and SGI Score Sensitivity Analysis
Catalyst Pharmaceuticals, Inc. - LMS-003
FAS Population (N=xxx)

| Statistic <sup>a</sup> | QMG Total Score | SGI Score |
|---|---|---|
| | | _ |
| P-value for Between-Treatment Difference in LS Means | XXX | XXX |

Source Program: xxxxxxx.sas

Source Listing: Data Listing 13, Data Listing 14

<sup>&</sup>lt;sup>a</sup> P-value based on conducting a randomization test by running the fixed effects linear model analysis on permuted treatment assignments. For each of the xxxx permutations, CFB was modeled as the response for each endpoint, with fixed effects terms for treatment and score at Baseline.

Table Creation Date: (DD-MMM-YYYY)

Page x of y

Table 25. CGI-I Scores Summary Statistics Catalyst Pharmaceuticals, Inc. - LMS-003 FAS Population (N=xxx)

| Treatment | Time Point | Mean | Std<br>Dev | n | Min | Max | Median | P-value <sup>a</sup> |
|---|---|---|---|---|---|---|---|---|
| Amifampridine | Day 4 | xxx | xxx | XXX | XXX | XXX | xxx | xxx |
| Placebo | Day 4 | xxx | XXX | xxx | xxx | xxx | xxx | |

Table Creation Date: (DD-MMM-YYYY)

Source Program: xxxxxxx.sas Source Listing: Data Listing 15

a P-value based on the Wilcoxon Rank Sum Test for treatment differences.
Page x of y

July 12, 2017

### Table 27. CGI-I Scores Summary Statistics by Dose Group Catalyst Pharmaceuticals, Inc. - LMS-003 FAS Population (N=xxx)

| | | | | | Std | | | | |
|---|---|---|---|---|---|---|---|---|---|
| Treatment | Dose Group | Time Point | Data Type | Mean | Dev | n | Min | Max | Median |
| Amifampridine | | | | | | | | | |
| | Low Dose (< 60mg/day) | Day 4 | RAW | XXX | XXX | XXX | XXX | XXX | XXX |
| | High Dose (> 60mg/day) | Day 4 | RAW | XXX | XXX | XXX | XXX | XXX | XXX |
| | All Doses | Day 4 | RAW | XXX | XXX | XXX | XXX | XXX | XXX |
| Placebo | | | | | | | | | |
| | Low Dose (< 60mg/day) | Day 4 | RAW | XXX | XXX | XXX | XXX | XXX | XXX |
| | High Dose ( $\geq$ 60mg/day) | Day 4 | RAW | XXX | XXX | XXX | XXX | XXX | XXX |
| | All Doses | Day 4 | RAW | XXX | XXX | XXX | XXX | XXX | XXX |

Table Creation Date: (DD-MMM-YYYY)

Source Program: xxxxxxx.sas Source Listing: Data Listing 15

Page x of y

Table 29. Number and Proportion of Subjects with  $\geq$  20% Increase in 3TUG Average Time Catalyst Pharmaceuticals, Inc. - LMS-003 FAS Population (N=xxx)

| Calculation | Amifampridine<br>(N=xxx) | Placebo<br>(N=xxx) | P-value <sup>a</sup> |
|---|---|---|---|
| Denominator Based on Subjects Who Completed Day 0 3TUG | xxx/xxx (xxx) | xxx/xxx (xxx) | xxx |
| Denominator Based on Subjects Who Completed Day 0 and Day 4 3TUG | xxx/xxx (xxx) | xxx/xxx (xxx) | xxx |

Table Creation Date: (DD-MMM-YYYY) Source Program: xxxxxxx.sas Source Listing: Data Listing 16

<sup>&</sup>lt;sup>a</sup> P-value based on a two-sided Fisher's Exact Test of difference in treatment proportions.

Page x of y

Table 31. Number and Proportion of Subjects with  $\geq$  20% Increase in 3TUG Average Time by Dose Group Catalyst Pharmaceuticals, Inc. - LMS-003 FAS Population (N=xxx)

Low Dose(< 60mg/day)

High Dose(≥ 60mg/day)

| Calculation | Amifampridine (N=xxx) | Placebo (N=xxx) | Amifampridine (N=xxx) | Placebo (N=xxx) |
|---|---|---|---|---|
| Denominator Based on Subjects Who<br>Completed Day 0 3TUG | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |
| Denominator Based on Subjects Who<br>Completed Day 0 and Day 4 3TUG | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |

Table Creation Date: (DD-MMM-YYYY)

Source Program: xxxxxxx.sas Source Listing: Data Listing 16

Page x of y

Table 33. Summary of Patient Most Bothersome Symptom Catalyst Pharmaceuticals, Inc. - LMS-003 FAS Population (N=xxx)

| | | | | Std | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| Treatment | Time Point <sup>a</sup> | Data Type <sup>b</sup> | Mean | Dev | n | Min | Max | Median | P-value <sup>c</sup> |
| Amifampridine | Day 0 (Baseline) | RAW | xxx | xxx | xxx | xxx | XXX | XXX | |
| | Post-Baseline | RAW | XXX | XXX | XXX | XXX | XXX | xxx | |
| | | CFB | XXX | XXX | XXX | XXX | XXX | XXX | xxxx |
| Placebo | Day 0 (Baseline) | RAW | xxx | xxx | XXX | xxx | xxx | xxx | |
| | Post-Baseline | RAW | XXX | XXX | XXX | XXX | XXX | XXX | |
| | | CFB | XXX | XXX | xxx | XXX | XXX | XXX | |

Table Creation Date: (DD-MMM-YYYY)

Source Program: xxxxxxx.sas Source Listing: Data Listing 17

<sup>&</sup>lt;sup>a</sup> The post-treatment result will be the result obtained on Day 4, unless the subject discontinued treatment early, in which case the post-treatment result may be obtained at an earlier time point.

b RAW = observed data entered in the database; CFB = change from baseline.

<sup>&</sup>lt;sup>c</sup> P-value based on the Wilcoxon Rank Sum Test for treatment differences in CFB results.

Page x of y

Table 35. Summary of Patient Most Bothersome Symptom by Dose Group
Catalyst Pharmaceuticals, Inc. - LMS-003
FAS Population (N=xxx)

| | | | | | Std | | | | |
|---|---|---|---|---|---|---|---|---|---|
| Treatment | Dose Group | Time Point <sup>a</sup> | Data Type <sup>b</sup> | Mean | Dev | n | Min | Max | Median |
| Amifampridine | | | | | | | | | |
| | Low Dose (< 60mg/day) | Day 0 (Baseline) | RAW | XXX | XXX | XXX | XXX | XXX | XXX |
| | | Post-Baseline | RAW | XXX | XXX | XXX | XXX | XXX | XXX |
| | | | CFB | XXX | XXX | XXX | XXX | XXX | XXX |
| | High Dose (> 60mg/day) | Day 0 (Baseline) | RAW | XXX | XXX | XXX | XXX | XXX | XXX |
| | | Post-Baseline | RAW | XXX | XXX | XXX | XXX | XXX | XXX |
| | | | CFB | XXX | XXX | XXX | XXX | XXX | XXX |
| | All Doses | Day 0 (Baseline) | RAW | XXX | XXX | XXX | XXX | XXX | XXX |
| | | Post-Baseline | RAW | XXX | XXX | XXX | XXX | XXX | XXX |
| | | | CFB | XXX | XXX | XXX | XXX | XXX | XXX |
| Placebo | | | | | | | | | |
| | Low Dose (< 60mg/day) | Day 0 (Baseline) | RAW | XXX | XXX | XXX | XXX | XXX | XXX |
| | | Post-Baseline | RAW | XXX | XXX | XXX | XXX | XXX | XXX |
| | | | CFB | XXX | XXX | XXX | XXX | XXX | XXX |
| | High Dose (> 60mg/day) | Day 0 (Baseline) | RAW | XXX | XXX | XXX | XXX | XXX | XXX |
| | | Post-Baseline | RAW | XXX | XXX | XXX | XXX | XXX | XXX |
| | | | CFB | XXX | XXX | XXX | XXX | XXX | XXX |
| | All Doses | Day 0 (Baseline) | RAW | XXX | XXX | XXX | XXX | XXX | XXX |
| | | Post-Baseline | RAW | XXX | XXX | XXX | XXX | XXX | XXX |
| | | | CFB | XXX | XXX | XXX | XXX | XXX | XXX |

Table Creation Date: (DD-MMM-YYYY)
Source Program: xxxxxxx.sas

Source Listing: Data Listing 17

<sup>&</sup>lt;sup>a</sup> The post-treatment result will be the result obtained on Day 4, unless the subject discontinued treatment early, in which case the post-treatment result may be obtained at an earlier time point.

b RAW = observed data entered in the database; CFB = change from baseline.

Page x of y

Table 37. QMG Total Score Summary Statistics by Limb Domain and Time Point Catalyst Pharmaceuticals, Inc. - LMS-003 FAS Population (N=xxx)

| | | | | | Std | | | | |
|---|---|---|---|---|---|---|---|---|---|
| Limb Domain | Treatment | Time Point <sup>a</sup> | Data Type <sup>b</sup> | Mean | Dev | n | Min | Max | Median |
| Left Arm | Amifampridine | Day 0 | RAW | xxx | xxx | xxx | XXX | XXX | xxx |
| Here min | imitampitatio | (Baseline) | 14111 | 212121 | 212121 | 212121 | 212121 | 212121 | 717171 |
| | | Post-Baseline | RAW | XXX | XXX | XXX | XXX | XXX | XXX |
| | | | CFB | XXX | XXX | XXX | XXX | XXX | xxx |
| | Placebo | D 0 | Data | | | | | | |
| | Placedo | Day 0<br>(Baseline) | RAW | XXX | XXX | XXX | XXX | XXX | XXX |
| | | Post-Baseline | RAW | XXX | XXX | XXX | XXX | XXX | XXX |
| | | | CFB | XXX | XXX | XXX | XXX | XXX | XXX |
| Right Arm | Amifampridine | Day 0 | RAW | xxx | xxx | xxx | xxx | xxx | XXX |
| 1119110 111111 | 11M11amp11aine | (Baseline) | 14111 | ***** | ***** | ***** | | | |
| | | Post-Baseline | RAW | XXX | XXX | XXX | XXX | XXX | xxx |
| | | | CFB | XXX | xxx | XXX | XXX | xxx | XXX |
| | Placebo | Day 0 | RAW | xxx | xxx | xxx | xxx | xxx | XXX |
| | 1140020 | (Baseline) | 14111 | ***** | ***** | ***** | | | |
| | | Post-Baseline | RAW | XXX | XXX | XXX | XXX | XXX | xxx |
| | | | CFB | XXX | XXX | XXX | XXX | XXX | XXX |
| Left Leg | Amifampridine | Day 0 | RAW | XXX | XXX | XXX | XXX | XXX | XXX |
| | | (Baseline) | | | | | | | |
| | | Post-Baseline | RAW | XXX | XXX | XXX | XXX | XXX | XXX |
| | | | CFB | XXX | XXX | XXX | XXX | XXX | XXX |
| | Placebo | Day 0 | RAW | XXX | XXX | XXX | XXX | XXX | xxx |
| | | (Baseline) | | | | | | | |
| | | Post-Baseline | RAW | XXX | XXX | XXX | XXX | XXX | XXX |
| | | | CFB | XXX | XXX | XXX | XXX | XXX | XXX |

Page x of y

# Table 37 (cont.). QMG Total Score Summary Statistics by Limb Domain and Time Point Catalyst Pharmaceuticals, Inc. - LMS-003 FAS Population (N=xxx)

| | | | | | Std | | | | |
|---|---|---|---|---|---|---|---|---|---|
| Limb Domain | Treatment | Time Point <sup>a</sup> | Data Type <sup>b</sup> | Mean | Dev | n | Min | Max | Median |
| Right Leg | Amifampridine | Day 0<br>(Baseline) | RAW | XXX | XXX | XXX | XXX | XXX | XXX |
| | | Post-Baseline | RAW | XXX | XXX | XXX | XXX | XXX | XXX |
| | | | CFB | XXX | XXX | XXX | XXX | XXX | XXX |
| | Placebo | Day 0<br>(Baseline) | RAW | xxx | xxx | xxx | XXX | XXX | XXX |
| | | Post-Baseline | RAW | XXX | XXX | XXX | XXX | XXX | XXX |
| | | | CFB | XXX | XXX | XXX | xxx | XXX | XXX |
| Total of Region Scores | Amifampridine | Day 0<br>(Baseline) | RAW | XXX | xxx | xxx | xxx | xxx | XXX |
| | | Post-Baseline | RAW | XXX | XXX | XXX | XXX | XXX | XXX |
| | | | CFB | XXX | XXX | XXX | XXX | XXX | XXX |
| | Placebo | Day 0<br>(Baseline) | RAW | xxx | xxx | xxx | xxx | xxx | XXX |
| | | Post-Baseline | RAW | XXX | XXX | XXX | XXX | XXX | XXX |
| | | | CFB | XXX | XXX | XXX | XXX | XXX | XXX |

Table Creation Date: (DD-MMM-YYYY)

Source Program: xxxxxxx.sas Source Listing: Data Listing 14

<sup>&</sup>lt;sup>a</sup> The post-treatment result will be the result obtained on Day 4, unless the subject discontinued treatment early, in which case the post-treatment result may be obtained at an earlier time point.

b RAW = observed data entered in the database; CFB = change from baseline.

Page x of y

Table 39. Limb Domain Specific QMG Total Score CFB Analysis
Catalyst Pharmaceuticals, Inc. - LMS-003
FAS Population (N=xxx)

| Limb Domain | Statistic <sup>a</sup> | Amifampridine | Placebo |
|---|---|---|---|
| Left Arm Outstretched | n | XXX | XXX |
| | Least Squares (LS) Mean of Change from Baseline (CFB) | XXX | XXX |
| | Between-Treatment Difference in LS Means | XXX | |
| | 95% CI for Between-Treatment Difference in LS Means | (xxx, xxx) | |
| | P-value for Between-Treatment Difference in LS Means | XXX | |
| Right Arm Outstretched | n | XXX | XXX |
| | Least Squares (LS) Mean of Change from Baseline (CFB) | XXX | xxx |
| | Between-Treatment Difference in LS Means | XXX | |
| | 95% CI for Between-Treatment Difference in LS Means | (xxx, xxx) | |
| | P-value for Between-Treatment Difference in LS Means | XXX | |
| Left Leg Outstretched | n | XXX | XXX |
| | Least Squares (LS) Mean of Change from Baseline (CFB) | XXX | xxx |
| | Between-Treatment Difference in LS Means | XXX | |
| | 95% CI for Between-Treatment Difference in LS Means | (xxx, xxx) | |
| | P-value for Between-Treatment Difference in LS Means | XXX | |
| Right Leg Outstretched | n | XXX | XXX |
| | Least Squares (LS) Mean of Change from Baseline (CFB) | XXX | xxx |
| | Between-Treatment Difference in LS Means | XXX | |
| | 95% CI for Between-Treatment Difference in LS Means | (xxx, xxx) | |
| | P-value for Between-Treatment Difference in LS Means | XXX | |
| Total of Regions <sup>b</sup> | n | XXX | XXX |
| | Least Squares (LS) Mean of Change from Baseline (CFB) | XXX | xxx |
| | Between-Treatment Difference in LS Means | xxx | |
| | 95% CI for Between-Treatment Difference in LS Means | (xxx, xxx) | |
| | P-value for Between-Treatment Difference in LS Means | XXX | |

<sup>&</sup>lt;sup>a</sup> CFB for QMG score was modeled as the response, with fixed effects terms for treatment and QMG at Baseline.

Table Creation Date: (DD-MMM-YYYY)

xxxxxx.sas

Source Listing: Data Listing 14

 $<sup>^{\</sup>mbox{\scriptsize b}}$  Total is the CFB of the sum of the four regions listed above.

Page x of y

Table 41. Number and Percent of Subjects with Treatment Emergent Adverse Events
Catalyst Pharmaceuticals, Inc. - LMS-003
Safety Population (N=xxx)

| Adverse Event Categorya: | Amifampridine (N=xxx) | Placebo<br>(N=xxx) | Overall<br>(N=xxx) |
|---|---|---|---|
| Total Number of Treatment Emergent Adverse Events (TEAEs) | xxx | xxx | xxx |
| Subjects with at Least One TEAE | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |
| System Organ Class 1<br>Preferred Term 1 | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |
| Preferred Term 2 | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |
| System Organ Class 2 | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |
| Preferred Term 1 | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |
| Preferred Term 2 | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |

Table Creation Date: (DD-MMM-YYYY) Source Program: xxxxxxx.sas Source Listing: Data Listing 8

<sup>&</sup>lt;sup>a</sup> Adverse events coded with MedDRA Coding Dictionary Version XXX.

Page x of y

Table 42. Number and Percent of Subjects with Treatment Emergent Adverse Events by Dose Level

Catalyst Pharmaceuticals, Inc. - LMS-003

Safety Population (N=xxx)

| | Amifampridine | | | Placebo | | |
|---|---|---|---|---|---|---|
| Adverse Event Categorya: | Low Dose<br>(N=xxx) | High Dose<br>(N=xxx) | All Doses<br>(N=xxx) | Low Dose (N=xxx) | High Dose<br>(N=xxx) | All Doses<br>(N=xxx) |
| Total Number of Treatment Emergent Adverse Events (TEAEs) | xxx | xxx | xxx | xxx | xxx | xxx |
| Subjects with at Least One TEAE | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |
| System Organ Class 1 Preferred Term 1 | xxx (xxx%)<br>xxx (xxx%) | xxx (xxx%)<br>xxx (xxx%) | xxx (xxx%)<br>xxx (xxx%) | xxx (xxx%)<br>xxx (xxx%) | xxx (xxx%)<br>xxx (xxx%) | xxx (xxx%)<br>xxx (xxx%) |
| Preferred Term 2 System Organ Class 2 | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%)<br>xxx (xxx%) | xxx (xxx%) xxx (xxx%) | xxx (xxx%) |
| Preferred Term 1 Preferred Term 2 | xxx (xxx%)<br>xxx (xxx%) | xxx (xxx%)<br>xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |

Table Creation Date: (DD-MMM-YYYY)

Source Program: xxxxxxx.sas Source Listing: Data Listing 8

a Adverse events coded with MedDRA Coding Dictionary Version XXX.

Page x of y

Table 43. Summary of Treatment Emergent Adverse Events Catalyst Pharmaceuticals, Inc. - LMS-003

Safety Population (N=xxxx)

| | Amifampridine (N=xxx) | Placebo<br>(N=xxx) | Overall (N=xxx) |
|---|---|---|---|
| Subjects with at Least One Treatment Emergent Adverse Event (TEAE) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |
| Maximum TEAE Severity Grade | | | |
| Mild (Grade 1) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |
| Moderate (Grade 2) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |
| Severe (Grade 3) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |
| Life-threatening (Grade 4) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |
| Death (Grade 5) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |
| Highest Relationship of TEAE to Treatment | | | |
| Not Related | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |
| Possibly | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |
| Probably | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |
| Subjects with at Least One Serious TEAE | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |

Table Creation Date: (DD-MMM-YYYY)

Source Program: xxxxxxx.sas Source Listing: Data Listing 8

Page x of y

Table 44. Number and Percent of Subjects with Serious Treatment Emergent Adverse Events

Catalyst Pharmaceuticals, Inc. - LMS-003

Safety Population (N=xxx)

| Adverse Event Category <sup>a</sup> : | Amifampridine (N=xxx) | Placebo<br>(N=xxx) | Overall (N=xxx) |
|---|---|---|---|
| Total Number of Serious Treatment Emergent<br>Adverse Events (TESAEs) | xxx | xxx | xxx |
| Subjects with at Least One TESAE | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |
| System Organ Class 1 Preferred Term 1 Preferred Term 2 | xxx (xxx%)<br>xxx (xxx%)<br>xxx (xxx%) | xxx (xxx%)<br>xxx (xxx%) | xxx (xxx%)<br>xxx (xxx%)<br>xxx (xxx%) |
| System Organ Class 2 Preferred Term 1 | xxx (xxx%)<br>xxx (xxx%) | xxx (xxx%)<br>xxx (xxx%) | xxx (xxx%) |
| Preferred Term 2 | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |

Table Creation Date: (DD-MMM-YYYY) Source Program: xxxxxxx.sas Source Listing: Data Listing 8

a Adverse events coded with MedDRA Coding Dictionary Version XXX.

Page x of y

Table 45. Number and Percent of Subjects with Treatment Emergent Adverse Events by Relationship to Treatment
Catalyst Pharmaceuticals, Inc. - LMS-003
Safety Population (N=xxx)

| | | Amifampridine<br>(N=xxx) | | Placebo<br>(N=xxx) | | |
|---|---|---|---|---|---|---|
| Adverse Event Categorya: | Not Related | Possibly | Probably | Not Related | Possibly | Probably |
| Total Number of Treatment Emergent Adverse Events (TEAEs) | xxx | xxx | xxx | xxx | xxx | xxx |
| Subjects with at Least One TEAE | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |
| System Organ Class 1 Preferred Term 1 Preferred Term 2 | xxx (xxx%)<br>xxx (xxx%)<br>xxx (xxx%) | xxx (xxx%)<br>xxx (xxx%)<br>xxx (xxx%) | xxx (xxx%)<br>xxx (xxx%)<br>xxx (xxx%) | xxx (xxx%)<br>xxx (xxx%)<br>xxx (xxx%) | xxx (xxx%)<br>xxx (xxx%)<br>xxx (xxx%) | xxx (xxx%)<br>xxx (xxx%) |
| System Organ Class 2 Preferred Term 1 Preferred Term 2 | xxx (xxx%) xxx (xxx%) | xxx (xxx%)<br>xxx (xxx%)<br>xxx (xxx%) | xxx (xxx%)<br>xxx (xxx%)<br>xxx (xxx%) | xxx (xxx%)<br>xxx (xxx%)<br>xxx (xxx%) | xxx (xxx%)<br>xxx (xxx%)<br>xxx (xxx%) | xxx (xxx%)<br>xxx (xxx%) |

Table Creation Date: (DD-MMM-YYYY)

Source Program: xxxxxxx.sas Source Listing: Data Listing 8

<sup>&</sup>lt;sup>a</sup> Adverse events coded with MedDRA Coding Dictionary Version XXX.

Page x of y

Table 46. Number and Percent of Subjects with Treatment Emergent Adverse Events by Severity Grade Catalyst Pharmaceuticals, Inc. - LMS-003 Safety Population (N=xxx)

Part 1 of 2

#### Amifampridine (N=xxx)Adverse Event Categorya: Grade 1 Grade 2 Grade 3 Grade 4 Grade 5 Total Number of Treatment Emergent XXX XXX XXX XXX XXX Adverse Events (TEAEs) Subjects with at Least One TEAE xxx (xxx%) xxx (xxx%) xxx (xxx%) xxx (xxx%) xxx (xxx%) System Organ Class 1 XXX (XXX%) XXX (XXX%) XXX (XXX%) XXX (XXX%) Preferred Term 1 XXX (XXX%) XXX (XXX%) XXX (XXX%) XXX (XXX%) XXX (XXX%) Preferred Term 2 XXX (XXX%) XXX (XXX%) XXX (XXX%) XXX (XXX%) XXX (XXX%) xxx (xxx%) xxx (xxx%) xxx (xxx%) xxx (xxx%) xxx (xxx%) System Organ Class 2 Preferred Term 1 XXX (XXX%) XXX (XXX%) XXX (XXX%) XXX (XXX%) XXX (XXX%) Preferred Term 2 XXX (XXX%) XXX (XXX%) XXX (XXX%) XXX (XXX%) XXX (XXX%)

Table Creation Date: (DD-MMM-YYYY)

Source Program: xxxxxxx.sas Source Listing: Data Listing 8

Version 1.0

a Adverse events coded with MedDRA Coding Dictionary Version XXX.

Page x of y

# Table 46 (cont.). Number and Percent of Subjects with Treatment Emergent Adverse Events by Severity Grade Catalyst Pharmaceuticals, Inc. - LMS-003 Safety Population (N=xxx)

Part 2 of 2

Placebo (N=xxx)Adverse Event Categorya: Grade 1 Grade 2 Grade 3 Grade 4 Grade 5 Total Number of Treatment Emergent XXX XXXXXX XXX XXXAdverse Events (TEAEs) Subjects with at Least One TEAE xxx (xxx%) xxx (xxx%) xxx (xxx%) xxx (xxx%) xxx (xxx%) System Organ Class 1 XXX (XXX%) XXX (XXX%) XXX (XXX%) XXX (XXX%) Preferred Term 1 XXX (XXX%) XXX (XXX%) XXX (XXX%) XXX (XXX%) XXX (XXX%) Preferred Term 2 xxx (xxx%) xxx (xxx%) xxx (xxx%) xxx (xxx%) xxx (xxx%) System Organ Class 2 XXX (XXX%) XXX (XXX%) XXX (XXX%) XXX (XXX%) Preferred Term 1 XXX (XXX%) XXX (XXX%) XXX (XXX%) XXX (XXX%) XXX (XXX%) Preferred Term 2 xxx (xxx%) xxx (xxx%) xxx (xxx%) xxx (xxx%) xxx (xxx%)

Table Creation Date: (DD-MMM-YYYY)

Source Program: xxxxxxx.sas
Source Listing: Data Listing 8

a Adverse events coded with MedDRA Coding Dictionary Version XXX.

Page x of y

Table 47. Vital Signs Summary Statistics Catalyst Pharmaceuticals, Inc. - LMS-003 Safety Population (N=xxx)

| Treatment | Vital Sign Parameter (units) | Visit | Data Typeª | Mean | Std<br>Dev | n | Min | Max | Median |
|---|---|---|---|---|---|---|---|---|---|
| Amifampridine | xxxxxxxxx (xxx) | Screening (Baseline) | RAW | XXX | XXX | XXX | xxx | xxx | xxx |
| | | Day X | RAW | XXX | XXX | XXX | XXX | XXX | XXX |
| | | | CFB | XXX | XXX | XXX | XXX | XXX | XXX |
| Placebo | xxxxxxxxx (xxx) | Screening (Baseline) | RAW | xxx | XXX | xxx | xxx | xxx | XXX |
| | | Day X | RAW | XXX | XXX | XXX | XXX | XXX | XXX |
| | | | CFB | XXX | XXX | XXX | XXX | XXX | XXX |

Table Creation Date: (DD-MMM-YYYY)
Source Program: xxxxxxx.sas

Source Program: xxxxxxx.sas Source Listing: Data Listing 10

<sup>&</sup>lt;sup>a</sup> RAW = observed data recorded in database; CFB = change from baseline

Page x of y

| Concomitant Medication Category <sup>a,b</sup> | Amifampridine<br>(N=xxx) | Placebo<br>(N=xxx) | Overall (N=xxx) |
|---|---|---|---|
| ATC Level 3 Term | xxxx (xxxx%) | xxxx (xxxx%) | xxxx (xxxx%) |
| WHO Preferred Term | xxxx (xxxx%) | xxxx (xxxx%) | xxxx (xxxx%) |
| WHO Preferred Term | xxxx (xxxx%) | xxxx (xxxx%) | xxxx (xxxx%) |
| ATC Level 3 Term | xxxx (xxxx%) | xxxx (xxxx%) | xxxx (xxxx%) |
| WHO Preferred Term | xxxx (xxxx%) | xxxx (xxxx%) | xxxx (xxxx%) |
| WHO Preferred Term | xxxx (xxxx%) | xxxx (xxxx%) | xxxx (xxxx%) |

Table Creation Date: (DD-MMM-YYYY)
Source Program: xxxxxxx.sas

Source Listing: Data Listing 7

 $<sup>^{\</sup>mathrm{a}}$  Concomitant medications coded with WHO Coding Dictionary xxxxxxxxxxx.

b Concomitant medication categories will include anatomical therapeutic chemical (ATC) level 3 term followed by preferred term.

Page x of y

Data Listing 1. Subject Disposition Data Listing Catalyst Pharmaceuticals, Inc. - LMS-003

| Subject | | | | Date of | |
|---|---|---|---|---|---|
| | Treatment | No. | Disposition Status | Disposition | Withdrawal Reason |
| | XXXXXX | XXXX | XXXXXXXXXXXXXXXXXXXXX | XXXXXXXX | XXXXXXXXXXXXXXXXXXXXXXXXXXX |
| | XXXXXX | XXXX | XXXXXXXXXXXXXXXXXXXXX | XXXXXXXX | XXXXXXXXXXXXXXXXXXXXXXXXXXX |
| | XXXXXX | XXXX | xxxxxxxxxxxxxxxxx | xxxxxxxx | xxxxxxxxxxxxxxxxxxxxxxx |
| | XXXXXX | XXXX | XXXXXXXXXXXXXXXXXXXXXX | xxxxxxxx | xxxxxxxxxxxxxxxxxxxxxxxx |

Table Creation Date: (DD-MMM-YYYY)
Source Program: xxxxxxx.sas

Page x of y

Data Listing 2. Protocol Deviations Data Listing Catalyst Pharmaceuticals, Inc. - LMS-003 Safety Population (N=xxx)

| | Subject | Date of | | Deviation Major or |
|---|---|---|---|---|
| Treatment | No. | Deviation | Deviation Description | Minor |
| XXXXXX | XXXX | XXXXXX | XXXXXXXXXXXXXXXXXXXXXXXXXXX | XXXXXXXXX |
| XXXXXX | XXXX | XXXXXX | xxxxxxxxxxxxxxxxxxxxxxx | xxxxxxxxx |
| XXXXXX | XXXX | XXXXXX | xxxxxxxxxxxxxxxxxxxxxxx | xxxxxxxxx |
| XXXXXX | XXXX | XXXXXX | xxxxxxxxxxxxxxxxxxxxxxxx | xxxxxxxxx |

Table Creation Date: (DD-MMM-YYYY)
Source Program: xxxxxxx.sas

Page x of y

Data Listing 3. Demographics Data Listing Catalyst Pharmaceuticals, Inc. - LMS-003 Safety Population (N=xxx)

| | | Informed | | | | | |
|---|---|---|---|---|---|---|---|
| | Subject | Consent | Date of | Age | | | Screening |
| Treatment | No. | Date | Birth | (yrs) | Gender | Ethnicity | Weight (kg) |
| XXXXXX | XXXX | XXXXXX | XXXXXX | XXX | XXXXXX | XXXXXX | XXXXXX |

Table Creation Date: (DD-MMM-YYYY)

Page x of y

Data Listing 4. Subjects Excluded from FAS Population Data Listing Catalyst Pharmaceuticals, Inc. - LMS-003
Safety Population (N=xxx)

| Treatment | Subject No. | Reason for Exclusion |
|-----------|-------------|-----------------------------|
| XXXXXX | XXXX | xxxxxxxxxxxxxxxxxxxx |
| XXXXXX | XXXX | XXXXXXXXXXXXXXXXXXXXXXXXXXX |
| XXXXXX | XXXX | xxxxxxxxxxxxxxxxxxxxxxx |
| XXXXXX | XXXX | xxxxxxxxxxxxxxxxxxxxxxx |

Table Creation Date: (DD-MMM-YYYY)
Source Program: xxxxxxx.sas

Page x of y

Data Listing 5. Subjects Excluded from PP Population Data Listing Catalyst Pharmaceuticals, Inc. - LMS-003

All Enrolled Subjects (N=xxx)

| Treatment | Subject No. | Reason for Exclusion |
|-----------|-------------|----------------------------|
| XXXXXX | XXXX | XXXXXXXXXXXXXXXXXXXXXXXXXX |
| XXXXXX | XXXX | XXXXXXXXXXXXXXXXXXXXXXXXXX |
| XXXXXX | XXXX | xxxxxxxxxxxxxxxxxxxxxx |
| XXXXXX | XXXX | xxxxxxxxxxxxxxxxxxxxxxxx |

Table Creation Date: (DD-MMM-YYYY)
Source Program: xxxxxxxx.sas

Page x of y

Data Listing 6. Medical History Data Listing Catalyst Pharmaceuticals, Inc. - LMS-003 Safety Population (N=xxx)

MedDRA System Organ Classa/

| | Subject | MedDRA Preferred Term/ | a | |
|---|---|---|---|---|
| Treatment | No. | CRF Verbatim Term | Start Date | Ongoing? |
| XXXXXX | xxxx | ********** | xxxxxx | XXX |
| | | xxxxxxxxxxxxxxxxxxxxxxxxxxxxx | XXXXXXX | XXX |
| | | xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx | xxxxxxx | XXX |

 $<sup>^{\</sup>rm a}$  Medical history terms coded with MedDRA Coding Dictionary Version xxx. Table Creation Date: (DD-MMM-YYYY)

Page x of y

Data Listing 7. Prior and Concomitant Medications Data Listing Catalyst Pharmaceuticals, Inc. - LMS-003 Safety Population (N=xxx)

| Treatment | Subject<br>No. | Verbatim Drug Name/<br>Indication/<br>ATC Level 3 Term | Start<br>Date | Stop<br>Date | Route | Ongoing? |
|---|---|---|---|---|---|---|
| xxxxxx | xxxxxxx | ************************************** | xxxxxx | xxxxxx | xxxxx | xxxxx |
| xxxxxx | xxxxxxx | ************************************** | xxxxxx | xxxxxx | xxxxx | xxxxx |

WHO Preferred Terma/

Table Creation Date: (DD-MMM-YYYY)
Source Program: xxxxxxx.sas

a Concomitant medications coded with WHO Coding Dictionary xxxxxxxxx

Page x of y

Data Listing 8. Adverse Events Data Listing Catalyst Pharmaceuticals, Inc. - LMS-003 Safety Population (N=xxx)

| Treatment | Dose | Subject<br>No. | Start Date and Time/ End Date and Time | Treatment<br>Start Date | MedDRA System<br>Organ Class <sup>a</sup> /<br>MedDRA Preferred<br>Term/<br>CRF Verbatim Term | Severity<br>Grade | Relation to<br>Treatment | Serious? | Outcome |
|---|---|---|---|---|---|---|---|---|---|
| xxxxx | xxxxx | xxxxxxxx | xxxxxx<br>xxxxxx/<br>xxxxxx<br>xxxxxx | xxxxxx | ************************************** | xxxxxxx | xxxxxxx | xxx | xxxxxxx |
| xxxxx | xxxxx | xxxxxxxx | xxxxxxx<br>xxxxxxx/<br>xxxxxxx<br>xxxxxxx | xxxxxx | ************************************** | xxxxxxx | xxxxxxx | xxx | xxxxxxx |

Table Creation Date: (DD-MMM-YYYY)

a Adverse events coded with MedDRA Coding Dictionary Version xxx.

Page x of y

Data Listing 9. Physical Exam Data Listing Catalyst Pharmaceuticals, Inc. - LMS-003 Safety Population (N=xxx)

| Treatment | Subject<br>No. | Visit | Date<br>Conducted | Body System | Result | Abnormality |
|---|---|---|---|---|---|---|
| XXXXXX | XXXX | XXXXXXX | xxxxxx | xxxxxxx | xxxxxxx | xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx |
| | | | | XXXXXXX | xxxxxxxx | xxxxxxxxxxxxxxxxxxxxxxxxxxxxx |
| | | | | XXXXXXX | xxxxxxxx | xxxxxxxxxxxxxxxxxxxxxxxxxxxxx |
| | | | | XXXXXXX | xxxxxxxx | xxxxxxxxxxxxxxxxxxxxxxxxxxxxx |
| | | | | xxxxxxx | xxxxxxxx | xxxxxxxxxxxxxxxxxxxxxxxxxxxxx |
| | | | | XXXXXXX | xxxxxxxx | xxxxxxxxxxxxxxxxxxxxxxxxxxxxx |
| | | | | XXXXXXX | xxxxxxxx | xxxxxxxxxxxxxxxxxxxxxxxxxxxxx |
| | | | | XXXXXXX | xxxxxxxx | xxxxxxxxxxxxxxxxxxxxxxxxxxxxx |
| | | | | xxxxxxx | xxxxxxxx | xxxxxxxxxxxxxxxxxxxxxxxxxxxxx |
| | | | | XXXXXXX | xxxxxxx | xxxxxxxxxxxxxxxxxxxxxxxxxxxxxx |

Table Creation Date: (DD-MMM-YYYY)

Page x of y

Data Listing 10. Vital Signs Data Listing Catalyst Pharmaceuticals, Inc. - LMS-003 Safety Population (N=xxx)

| | | | | | | Systolic<br>Blood | Diastolic<br>Blood | Heart |
|---|---|---|---|---|---|---|---|---|
| | Subject | | | | Temp. | Pressure | Pressure | Rate |
| Treatment | No. | Visit | Date | Time | (°F) | (mmHg) | (mmHg) | (bpm) |
| XXXXXX | XXXX | XXXXXXX | XXXXXXX | XXXXX | XXX | XXX | XXX | XXX |
| | | | | XXXXX | XXX | XXX | XXX | XXX |
| | | | | XXXXX | XXX | XXX | XXX | XXX |
| XXXXXX | XXXX | XXXXXXX | XXXXXXX | XXXXX | XXX | XXX | XXX | XXX |
| | | | | XXXXX | XXX | XXX | XXX | XXX |
| | | | | XXXXX | XXX | XXX | XXX | XXX |

Table Creation Date: (DD-MMM-YYYY)

Page x of y

Data Listing 11. Study Drug Administration Data Listing Catalyst Pharmaceuticals, Inc. - LMS-003

Safety Population (N=xxx)

| Treatment | Subject<br>No. | Treatment<br>Start<br>Date | Treatment<br>End Date | Treatment<br>Duration<br>(Days) | Tablets<br>Consumed | Dose Group<br>(Low or High) <sup>a</sup> | Tablets<br>Prescribed <sup>b</sup> | Compliance (%)° |
|---|---|---|---|---|---|---|---|---|
| XXXXXX | XXXX | XXXXXX | XXXXXX | xxx | xxx | XXX | xxx | XXX |
| xxxxxx | xxxx | xxxxxx | xxxxxx | xxx | xxx | XXX | xxx | xxx |

Table Creation Date: (DD-MMM-YYYY)

 $<sup>^{</sup>a}$  Low dose group is < 60mg/day and high dose group is  $^{>}$  60mg/day, based on prescribed tablets.

b Number of tablets prescribed is computed as the duration times the number of tablets to have been taken daily.

 $<sup>^{\</sup>circ}$  Compliance is computed as 100%\*(number of tablets consumed)/(number of tables prescribed).

Page x of y

Data Listing 12. SGI Data Listing Catalyst Pharmaceuticals, Inc. - LMS-003 Safety Population (N=xxx)

| Subject | | | Impression of Effects of Study Medication During |
|---|---|---|---|
| Treatment | No. | Visit | Preceding 3 Days on Physical Well Being <sup>a</sup> |
| xxxxxx | xxxx | xxxxxxx | xxxx |
| xxxxx | XXXX | xxxxxxx | XXXX |

Table Creation Date: (DD-MMM-YYYY)

a 1=Terrible; 2=Mostly Dissatisfied; 3=Mixed; 4=Partially Satisfied; 5=Mostly Satisfied; 6=Pleased; 7=Delighted.

Page x of y

## Data Listing 13. QMG Data Listing Catalyst Pharmaceuticals, Inc. - LMS-003 Safety Population (N=xxx)

| | Subject | | | |
|---|---|---|---|---|
| Treatment | No. | Visit | Item | Score |
| XXXXXX | XXXX | XXXXXXXX | Double Vision (Lateral Gaze) Sec. | XXXX |
| | | | Ptosis (Upward Gaze) Sec. | XXXX |
| | | | Facial Muscles | XXXX |
| | | | Swallowing 4oz. Water (1/2 cup) | XXXX |
| | | | Speech Following Counting Aloud From 1-50 (Onset of Dysarthria) | xxxx |
| | | | Right Arm Outstretched (90°, sitting) Sec. | XXXX |
| | | | Left Arm Outstretched (90°, sitting) Sec. | XXXX |
| | | | Forced Vital Capacity | xxxx |
| | | | Right Hand Grip (kg) | xxxx |
| | | | Left Hand Grip (kg) | xxxx |
| | | | Head, Lifted (45%, supine) Sec. | xxxx |
| | | | Right Leg Outstretched (45-50%, supine) Sec. | xxxx |
| | | | Left Leg Outstretched (45-50%, supine) Sec. | xxxx |
| | | | TOTAL | xxxx |

Table Creation Date: (DD-MMM-YYYY)

Page x of y

Data Listing 14. CGI-I Data Listing Catalyst Pharmaceuticals, Inc. - LMS-003 Safety Population (N=xxx)

| | Subject | | How Much Has Subject's Condition |
|-----------|---------|---------|----------------------------------|
| Treatment | No. | Visit | Changed Since Day 0?a |
| xxxxxx | xxxx | xxxxxxx | xxxx |
| xxxxxx | xxxx | xxxxxxx | XXXX |

<sup>&</sup>lt;sup>a</sup> 1=Very Much Improved; 2=Much Improved; 3=Minimally Improved; 4=No Change; 5=Minimally Worse; 6=Much Worse; 7=Very Much Worse. Table Creation Date: (DD-MMM-YYYY)

Page x of y

### Data Listing 15. 3TUG Data Listing Catalyst Pharmaceuticals, Inc. - LMS-003 Safety Population (N=xxx)

| | Subject | | Time | % Increase from |
|-----------|---------|------------------|-------|-----------------|
| Treatment | No. | Visit | (Sec) | Baseline |
| xxxxxx | xxxx | Day 0 (Baseline) | xxxx | |
| xxxxxx | XXXX | xxxxxxx | xxxx | xxxx |

Table Creation Date: (DD-MMM-YYYY)

Page x of y

Data Listing 16. Patient Most Bothersome Symptom Data Listing Catalyst Pharmaceuticals, Inc. - LMS-003 Safety Population (N=xxx)

| | Subject | | Rating of Most Bothersome | Rating of Most Bothersome Symptom During the Last 24 Hours After |
|---|---|---|---|---|
| Treatment No. Visit | | | Symptom Before Treatment <sup>a</sup> | Treatment with Study Medication |
| xxxxxx | XXXX | xxxxxxx | xxxx | xxxx |
| xxxxxx | xxxx | xxxxxxx | XXXX | xxxx |

Table Creation Date: (DD-MMM-YYYY)

a 0=Not At All Bothersome; 1=Bothered Me a Little; 2=Bothered Me Some; 3=Bothered Me a Lot.

 $<sup>^{\</sup>mathrm{a}}$  O=Not At All Bothersome; 1=Bothers Me a Little; 2=Bothers Me Some; 3=Bothers Me a Lot.

Page x of y

### Data Listing 17 - Subject Data Profile Catalyst Pharmaceuticals, Inc. Safety Population (N=xxx)

| Study Number: | : LMS-003 | Site: xxxxxxxxx | Subject ID: xxxxx | |
|---|---|---|---|---|
| Randomizatior<br>Age (yrs): xx | | Treatment: xxxxxx Gender: xxxxxx | Dose: xxxxxx<br>Ethnicity: xxxxxxx | Dose Group: xxx |
| Screening Wei | ight (kg): xxxx | | | |
| Endpoint Meas | surements | | | |
| паротис меаз | 3 dI ements | <del></del> | | |
| Subject Gener<br>Visit | ral Impression:<br>Date | Score | CFB | |
| Baseline | XX-XXX-XXXX | XXXXXX | | • |
| Day 4 | xx-xxx-xxxx | xxxxx | XXXXXX | |
| Ouantitative | Myasthenia Gravis | Scores | | |
| /isit | Date | Item | Score | CI |
| Baseline | xx-xxx-xxxx | Double vision | XXXXX | |
| | | Ptosis | xxxxx | - |
| | | Facial Muscles | xxxxx | - |
| | | Swallowing | xxxxx | |
| | | Speech following counting | from 1-50 xxxxx | |
| | | Right arm outstretched | xxxxx | |
| | | Left arm outstretched | xxxxx | |
| | | Forced vital capacity | xxxxx | |
| | | Right hand grip | xxxxx | |
| | | Left hand grip | xxxxx | |
| | | Head, lifted | xxxxx | |
| | | Right leg outstretched | XXXXX | |
| | | Left leg outstretched | XXXXX | |
| | | Limb total | XXXXX | |
| | | Total Score | XXXXX | |
| ay x | xx-xxx-xxx | Double vision | XXXXX | XXX |
| | | Ptosis | XXXXX | XXX |
| | | Facial Muscles | XXXXX | XXX |
| | | Swallowing | XXXXX | XXX |
| | | Speech following counting | from 1-50 xxxxx | XXX |
| | | Right arm outstretched | XXXXX | XXX |
| | | Left arm outstretched | XXXXX | XXX |
| | | Forced vital capacity | XXXXX | XXX |
| | | Right hand grip | XXXXX | XXX |
| | | Left hand grip | XXXXX | XXX |
| | | Head, lifted | XXXXX | XXX |
| | | Right leg outstretched | XXXXX | XXX |
| | | Left leg outstretched | xxxxx | XXX |
| | | Limb total | XXXXX | XXX |
| | | Total Score | XXXXX | XXX |
| Clinical Glob | oal Impression | xxxxxxx | | |
| l'riple Timed<br>Cime | Up and Go (3TUG) S Date | cores<br>Score | CFB | |
| Baseline | xx-xxx-xxxx | XXXX | | • |
| Day xxx | xx-xxx-xxxx | XXXX | XXXX | |
| Patient Most | Bothersome Symptom | | | |
| Time | Date | Score | CFB | |
| Baseline | xx-xxx-xxx | XXXX | | |

Page 70 of 71

Page x of y

### Data Listing 17 - Subject Data Profile Catalyst Pharmaceuticals, Inc. Safety Population (N=xxx)

| Study Number: LMS- | 003 | Site: xxxxxxxxx | Subject ID: xxxxx | |
|---|---|---|---|---|
| Laboratory Values<br>Visit | Date | Parameter (units) | Result | Abnormal Criterion |
| Baseline | XX-XXX-XXXX | xxxxxxxxxxxxxxxx | XXXX | |
| | | xxxxxxxxxxxxxxxxx | XXXX | |
| | | xxxxxxxxxxxxxxxxx | XXXX | |
| | | xxxxxxxxxxxxxxxxx | XXXX | |
| Day x | xx-xxx-xxxx | xxxxxxxxxxxxxxxxx | XXXX | |
| | | xxxxxxxxxxxxxxxxx | XXXX | |
| | | xxxxxxxxxxxxxxxx | XXXX | |
| | | xxxxxxxxxxxxxxxx | XXXX | |
| Vital Signs | | | | |
| Visit | Date | Parameter (units) | Result | Abnormal Criterion |
| Baseline | XX-XXX-XXXX | xxxxxxxxxxxxxxxxxxxxx | XXXX | |
| | XX-XXX-XXXX | xxxxxxxxxxxxxxxxxxx | XXXX | |
| | xx-xxx-xxxx | xxxxxxxxxxxxxxxxxxxxxxxx | XXXX | |
| Day x | xx-xxx-xxx | xxxxxxxxxxxxxxxxxxxxx | xxxx | |
| | xx-xxx-xxxx | xxxxxxxxxxxxxxxxxxxxxx | XXXX | |
| | xx-xxx-xxxx | xxxxxxxxxxxxxxxxxxx | xxxx | |
| Adverse Events <sup>a</sup><br>Event | | | | |
| (Preferred Term) | Date | System Organ Class | Severity | Treatment Related? |
| XXXXXXXXX | XX-XXX-XXXX | xxxxxxxxxxxxxxxxx | XXXX | XXXXXXXXX |
| XXXXXXXXXX | XX-XXX-XXXX | XXXXXXXXXXXXXXXXXXXXX | XXXX | XXXXXXXXX |
| XXXXXXXXXX | XX-XXX-XXXX | xxxxxxxxxxxxxxxxxx | XXXX | XXXXXXXXX |
| XXXXXXXXX | xx-xxx-xxxx | xxxxxxxxxxxxxxxxxx | XXXX | xxxxxxxxx |
| Prior and Concomit<br>Medication | ant Medications | d | | |
| (Preferred Term) | Dose | Start Date | Stop Date | |
| XXXXXXX | XXXXX | xx-xxx-xxxx | XX-XXX-XX | XXX |
| XXXXXXX | XXXXX | XX-XXX-XXXX | XX-XXX-XX | XXX |
| XXXXXXX | XXXXX | XX-XXX-XXXX | XX-XXX-XX | XXX |
| XXXXXXX | XXXXX | xx-xxx-xxxx | XX-XXX-XX | XXX |
| XXXXXXX | XXXXX | xx-xxx-xxxx | xx-xxx-xx | xxx |

Table Creation Date: (DD-MMM-YYYY)
Source Program: xxxxxxx.sas

### Table repeats per Subject beginning on a new page.

<sup>&</sup>lt;sup>a</sup> Adverse events coded with MedDRA Coding Dictionary Version xxx.

 $<sup>^{\</sup>rm b}$  Concomitant medications coded with WHO Coding Dictionary xxxxxxxx